CLINICAL TRIAL: NCT04581304
Title: The Use of Bio-Oss Collagen for Sinus Augmentation Using the Transcrestal Approach.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Hadar Zigdon MD, Rambam Health Care Campus, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0136-20-RMB CTIL
Record Dates: First submitted 2020-10-04; First posted 2020-10-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Bone Loss; Missing Teeth
MeSH Terms: conditions — Bone Diseases, Metabolic; Anodontia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-Oss Collagen (Experimental): Transcrestal approach sinus augmentation using Geistlich Bio-Oss Collagen®.
  Interventions: Device: Geistlich Bio-Oss® Collagen
- Bio-Oss Granules (Active Comparator): Transcrestal approach sinus augmentation using Geistlich Bio-Oss®.
  Interventions: Device: Geistlich Bio-Oss® Granules

INTERVENTIONS:
Device: Geistlich Bio-Oss® Collagen — Geistlich Bio-Oss® Collagen is intended to be used for filling bone defects and for bone augmentation.
  Arms: Bio-Oss Collagen
Device: Geistlich Bio-Oss® Granules — Geistlich Bio-Oss® Granules is intended to be used for filling bone defects and for bone augmentation.
  Arms: Bio-Oss Granules

SUMMARY:
To assess vertical bone height gain with Geistlich Bio-Oss Collagen used in conjunction with simultaneous implant installation in transcrestal approach sinus augmentation.

DETAILED DESCRIPTION:
One of the most common situations in the posterior maxilla is reduced alveolar bone height as a result of tooth extraction and the following bone remodeling process, and maxillary sinus pneumatization. Lack of alveolar bone volume may compromise dental implant installation. Maxillary sinus augmentation is considered a very predictable solution for implant installation in limited amount of bone in the posterior maxilla. In general, there are two main maxillary sinus augmentation methods: the lateral approach and the transcrestal. In both methods, the idea is to expend the alveolar ridge in vertical direction on the expense of the maxillary sinus. Sinus augmentation using the transcrestal approach is a well known procedure which is being use for over 40 years. As time goes by, implant dentistry is evolving and improving, there is a constant progress in this field including new bone substitutes materials.

Geistlich Bio-Oss® Collagen - can improve the results obtained by sinus augmentation using the transcrestal approach, by better ease of use for the operator which makes it easier for the operator and the patient.

Study hypothesis: The vertical bone height gained by using Geistlich Bio-Oss Collagen in transcrestal approach sinus augmentation will be comparable to using Bio-Oss Collagen, with greater operator satisfaction and less intra-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18.
* Patients with edentulous ridge maximal height of 8mm≥ beneath the maxillary sinus.
* Patients with edentulous ridge minimal height of 3mm≤ beneath the maxillary sinus.
* Patients who need single implant placement at the posterior maxilla.
* Signed, well filled and dated informed consent form.

Exclusion Criteria:

* Inability to complete or understand the informed consent process.
* Pregnant women.
* Lactating women.
* Patients who use medications that affect bone metabolism such as IV bisphosphonates.
* Heavy smokers.
* Patients with chronic/acute sinus infections

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2028-01-17 (Estimated)

PRIMARY OUTCOMES:
Vertical bone height. (mm)Changes in augmented bone after transcrestal approach sinus augmentation. | Pre op; immediately post-op, at 6 months and 3 years from second stage surgery.
  Measuring the changes in augmented bone volume after transcrestal approach sinus augmentation.

SECONDARY OUTCOMES:
Procedure time measurement. (min) | The procedure time measurement will start after flaps are elevated at pilot drilling (2.4mm diameter). and it will be stopped when the implant was inserted and insertion torque was assessed.
  To evaluate the time needed for transcrestal approach sinus augmentation using Bio-Oss collagen® and in the conventional way, using Bio-Oss granules.
Patients and operator satisfaction. (1-10 ruler scale) | At the suture removal visit - 14 days after procedure.
  To study operator and patients satisfaction using the 2 materials. They will be assessed by giving the patients questionnaires and satisfaction ruler using a 1-10 ruler scale.
Complications | During the procedure, During the follow up - 14 days, 6 months after intervention.
  Explore intra and post operative complications.
The success rate of osseointegrated implants. (%) | At 6 months and 3.5 years after intervention.
  The percentage of osseointegrated implants that were installed with simultaneous transcrestal approach sinus augmentation.- using Bio-Oss collagen®.

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Zigdon, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Dept. of Periodontology, Haifa, Israel